CLINICAL TRIAL: NCT04206579
Title: Oral 10% Dextrose Versus Sodium Dextrose Formula in Performance of Soccer Athlete. A Double-Blind Cross Over Randomized Controlled Trial
Brief Title: Oral Dextrose Formula in Performance of Soccer Athlete
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0611192027
Record Dates: First submitted 2019-12-12; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Athletes
Keywords: Oral Dextrose; Blood Sugar; Sprint Velocity; Athletes
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: the study involves two different groups with a cross-over design. Each participant will be given an oral formula according to the group allocation followed by outcome measurement. After the wash-out period, the formula will be switched and given to the participants, followed by outcome measurement
Who Masked: Participant, Investigator
Masking Description: Both packages of intervention have a similar dimension to ensure the participants are not recognizing the formula. The pharmacists are responsible for preparing the formula and given to the nurse prior to the intervention. Investigators are being masked during the whole intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10% Dextrose (Experimental): Oral 10% Dextrose
  Interventions: Drug: 10% Dextrose; Drug: Natrium Dextrose
- Natrium Dextrose (Experimental): Oral Natrium Dextrose
  Interventions: Drug: 10% Dextrose; Drug: Natrium Dextrose

INTERVENTIONS:
Drug: 10% Dextrose — A mixture of 150 cc dextrose 10% in oral formulation
  Other Names: Unavailable Information
Drug: Natrium Dextrose — A mixture of 150 cc dextrose 10% + 20 cc sodium in oral formulation
  Other Names: Unavailable Information

SUMMARY:
I. Title of Proposed Research Project Dextrose 10% Drink Increase Blood Sugar and Sprint Velocity Compared to Sodium Dextrose in Soccer Players

II. Specific Aims This study aims to evaluate the ergogenic effect in terms of blood sugar, VO2 max and sprint speed of dextrose 10% compared with sodium dextrose 10% in young male soccer players.

III. Background Sports drinks are designed to provide CHO, electrolytes, and fluids to the body, which are absorbed very fast from the small intestine. In other words, the period from ingestion until the CHO, electrolytes, and fluids reach the muscles, brain and so on, should be very short. This is the most important advantage of using sports drinks (Simulescu, Ilia, Macarie, & Merghes, 2019). Commercial sports drinks generally contain both of CHO and sodium; To the best of the investigator's knowledge, there is no trial in which compare the differential effect of solely dextrose supplementation versus sodium dextrose in soccer players in terms of BG concentration, VO2 max and sprint speed, which may give a new paradigm for the available ergogenic sports drink.

DETAILED DESCRIPTION:
Male academy soccer players, included in a trial, received two types of solutions (compound of 150 cc dextrose 10% + 20 mM sodium or single 150 cc dextrose 10%) interchangeably, separated within 120 minutes were completed in a counterbalanced, randomized, double-blind, crossover design. The study was approved by the Faculty of Medicine Hasanuddin University Research Ethics Committee. This trial was conducted at UNM Banta-Bantaeng, Makassar, Indonesia, from April 2019 to May 2019. All participants were within the last meal four hours prior to the test. Exclusion criteria were the use of amylase supplement, suffering from fever and diarrhea, using laxative agents within 24 h, consuming CHO absorption inhibitors, caffeine, creatinine, beta alanine, sodium bicarbonate supplement within 24 h, mean arterial pressure <65mmHg, knee or muscle injuries, history of diabetes mellitus and heart disease, going through ketogenic diet program, history of gastrointestinal surgery, and total body fat percentages > 30%.

Dietary intake was collected using two days food recall. BG were measured using portable glucometer (Aviva; Accucheck, Roche Diagnostics, Indiana, U.S.A), blood pressure were measured using aneroid sphygmomanometer (R1 shock-proof; Riester, Jungingen, Germany), heart rate were measured with wrist band pulse monitor (Bluetooth 4.0 wireless sport heart rate monitor WP290; Egoman, Shenzen, China), body weight, muscle, fat, water, metabolic rate were measured using body composition analyzer (BC-545N; Tanita, Tokyo, Japan), body height were measured using stadiometer (HR-200, Tanita, Tokyo, Japan), sprint speed were measured using digital stopwatch (S23589 S23589P1; Seiko, Tokyo, Japan) Participants were instructed to refrain from strenuous physical activity in the 2 days preceding trial sessions and recorded all food consumed in the 2 days before the trial. Food records subsequently were analyzed using professional German nutrition software (EBISpro, Nutrisurvey 2007). On arrival at the field, pre supplementation capillary blood samples were collected, and then all players run for 2x100 m and calculated the VO2max using Uth-Sorenen-Overgaard-Pedersen Formula and sprint speed was recorded. After doing the baseline measurement, each player waited for 15 minutes in order to consume either dextrose or sodium dextrose solution, and then waited for 15 minutes to had another subsequent capillary blood samples measurement. After that, the players run for 2x100 m, recorded the VO2max and sprint speed. The players remained in a rested state for 120 minutes as a crossover washed-out period, and then did the same protocol with different solution.

All data are expressed as mean ± SD unless otherwise stated, with 95% confidence interval, and significance was accepted at p < 0.05. Data were checked for normality as indicated by the Shapiro-Wilk test. Paired t tests were used to compare before and after condition in blood sugar, VO2max and sprint speed. Data was analysed using IBM SPSS Statistics software, version 25; IBM Corp., Chicago, IL. To interpret the magnitude of effect, Cohen's d effect sizes (±95% confidence limits) were estimated using a purpose built spreadsheet, with effect size thresholds set at <0.20, >0.50, and >0.80 for small, moderate, large, effects respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 18-23 years.
3. Soccer player
4. Last meal a maximum of 4 hours before
5. Willing and signed an agreement to participate in research.

Exclusion Criteria:

1. The use of amylase supplement
2. Suffering from fever and diarrhea
3. Using laxative agents within 24 h
4. Consuming CHO absorption inhibitors, Caffeine, creatinine, beta-alanine, sodium bicarbonate supplement within 24 h,
5. Mean arterial pressure <65mmHg
6. Knee or muscle injuries,
7. History of diabetes mellitus and heart disease
8. Going through the ketogenic diet program.
9. History of gastrointestinal surgery, and total body fat percentages > 30%.

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male at birth
Enrollment: 30 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | Blood Glucose Level at 15 minutes after intake
  Blood Glucose measured in capillary blood vessels

SECONDARY OUTCOMES:
Sprint Velocity | Sprint Velocity 30 minutes after intervention
  maximum sprint speed
Volume O2 maximum (VO2 Max) | VO2 10 minutes after sprint
  Maximum (MAX) volume (V) of oxygen (O2) an individual body in incremental exercise

CONTACTS AND LOCATIONS:
Overall Officials: Agussalim Bukhari, MD, Ph.D, Principal Investigator — Hasanuddin University
Locations (1):
- Makassar State University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared

REFERENCES:
- [Background] Achten J, Halson SL, Moseley L, Rayson MP, Casey A, Jeukendrup AE. Higher dietary carbohydrate content during intensified running training results in better maintenance of performance and mood state. J Appl Physiol (1985). 2004 Apr;96(4):1331-40. doi: 10.1152/japplphysiol.00973.2003. Epub 2003 Dec 5. PMID 14660506
- [Background] Afshar N, Safaei S, Nickerson DP, Hunter PJ, Suresh V. Computational Modeling of Glucose Uptake in the Enterocyte. Front Physiol. 2019 Apr 12;10:380. doi: 10.3389/fphys.2019.00380. eCollection 2019. PMID 31031632
- [Background] Amann M. Pulmonary system limitations to endurance exercise performance in humans. Exp Physiol. 2012 Mar;97(3):311-8. doi: 10.1113/expphysiol.2011.058800. Epub 2011 Nov 28. PMID 22125308
- [Background] Baker LB, Rollo I, Stein KW, Jeukendrup AE. Acute Effects of Carbohydrate Supplementation on Intermittent Sports Performance. Nutrients. 2015 Jul 14;7(7):5733-63. doi: 10.3390/nu7075249. PMID 26184303
- [Background] Bangsbo J, Iaia FM, Krustrup P. Metabolic response and fatigue in soccer. Int J Sports Physiol Perform. 2007 Jun;2(2):111-27. doi: 10.1123/ijspp.2.2.111. PMID 19124899
- [Background] Boyd CA, Parsons DS. Movements of monosaccharides between blood and tissues of vascularly perfused small intestine. J Physiol. 1979 Feb;287:371-91. doi: 10.1113/jphysiol.1979.sp012665. PMID 430421
- [Background] Burke LM, Meyer NL, Pearce J. National Nutritional Programs for the 2012 London Olympic Games: a systematic approach by three different countries. Nestle Nutr Inst Workshop Ser. 2013;76:103-20. doi: 10.1159/000350263. Epub 2013 Jul 25. PMID 23899758
- [Background] Dobbins RL, Greenway FL, Chen L, Liu Y, Breed SL, Andrews SM, Wald JA, Walker A, Smith CD. Selective sodium-dependent glucose transporter 1 inhibitors block glucose absorption and impair glucose-dependent insulinotropic peptide release. Am J Physiol Gastrointest Liver Physiol. 2015 Jun 1;308(11):G946-54. doi: 10.1152/ajpgi.00286.2014. Epub 2015 Mar 12. PMID 25767259
- [Background] Esposito BP, Breuer W, Sirankapracha P, Pootrakul P, Hershko C, Cabantchik ZI. Labile plasma iron in iron overload: redox activity and susceptibility to chelation. Blood. 2003 Oct 1;102(7):2670-7. doi: 10.1182/blood-2003-03-0807. Epub 2003 Jun 12. PMID 12805056
- [Background] F Alghannam, A. (2013). Physiology of Soccer: The Role of Nutrition in Performance. Journal of Novel Physiotherapies. https://doi.org/10.4172/2165-7025.s3-003
- [Background] Gabbett TJ, Mulvey MJ. Time-motion analysis of small-sided training games and competition in elite women soccer players. J Strength Cond Res. 2008 Mar;22(2):543-52. doi: 10.1519/JSC.0b013e3181635597. PMID 18550972
- [Background] Godek SF, Peduzzi C, Burkholder R, Condon S, Dorshimer G, Bartolozzi AR. Sweat rates, sweat sodium concentrations, and sodium losses in 3 groups of professional football players. J Athl Train. 2010 Jul-Aug;45(4):364-71. doi: 10.4085/1062-6050-45.4.364. PMID 20617911
- [Background] Hills SP, Russell M. Carbohydrates for Soccer: A Focus on Skilled Actions and Half-Time Practices. Nutrients. 2017 Dec 25;10(1):22. doi: 10.3390/nu10010022. PMID 29295583
- [Background] Jentjens RL, Achten J, Jeukendrup AE. High oxidation rates from combined carbohydrates ingested during exercise. Med Sci Sports Exerc. 2004 Sep;36(9):1551-8. doi: 10.1249/01.mss.0000139796.07843.1d. PMID 15354037
- [Background] Jeukendrup A. A step towards personalized sports nutrition: carbohydrate intake during exercise. Sports Med. 2014 May;44 Suppl 1(Suppl 1):S25-33. doi: 10.1007/s40279-014-0148-z. PMID 24791914
- [Background] Jeukendrup AE. Training the Gut for Athletes. Sports Med. 2017 Mar;47(Suppl 1):101-110. doi: 10.1007/s40279-017-0690-6. PMID 28332114
- [Background] Kellett GL. The facilitated component of intestinal glucose absorption. J Physiol. 2001 Mar 15;531(Pt 3):585-95. doi: 10.1111/j.1469-7793.2001.0585h.x. PMID 11251042
- [Background] Kellett GL, Brot-Laroche E. Apical GLUT2: a major pathway of intestinal sugar absorption. Diabetes. 2005 Oct;54(10):3056-62. doi: 10.2337/diabetes.54.10.3056. PMID 16186415
- [Background] Kellett GL, Brot-Laroche E, Mace OJ, Leturque A. Sugar absorption in the intestine: the role of GLUT2. Annu Rev Nutr. 2008;28:35-54. doi: 10.1146/annurev.nutr.28.061807.155518. PMID 18393659
- [Background] Kimmich GA, Randles J. Sodium-sugar coupling stoichiometry in chick intestinal cells. Am J Physiol. 1984 Jul;247(1 Pt 1):C74-82. doi: 10.1152/ajpcell.1984.247.1.C74. PMID 6331188
- [Background] Kingsley M, Penas-Ruiz C, Terry C, Russell M. Effects of carbohydrate-hydration strategies on glucose metabolism, sprint performance and hydration during a soccer match simulation in recreational players. J Sci Med Sport. 2014 Mar;17(2):239-43. doi: 10.1016/j.jsams.2013.04.010. Epub 2013 May 20. PMID 23702257
- [Background] Mace OJ, Affleck J, Patel N, Kellett GL. Sweet taste receptors in rat small intestine stimulate glucose absorption through apical GLUT2. J Physiol. 2007 Jul 1;582(Pt 1):379-92. doi: 10.1113/jphysiol.2007.130906. Epub 2007 May 10. PMID 17495045
- [Background] Mace OJ, Morgan EL, Affleck JA, Lister N, Kellett GL. Calcium absorption by Cav1.3 induces terminal web myosin II phosphorylation and apical GLUT2 insertion in rat intestine. J Physiol. 2007 Apr 15;580(Pt. 2):605-16. doi: 10.1113/jphysiol.2006.124784. Epub 2007 Feb 1. PMID 17272349
- [Background] MacLeod RJ, Hamilton JR. Volume regulation initiated by Na(+)-nutrient cotransport in isolated mammalian villus enterocytes. Am J Physiol. 1991 Jan;260(1 Pt 1):G26-33. doi: 10.1152/ajpgi.1991.260.1.G26. PMID 1702936
- [Background] Naftalin RJ. Does apical membrane GLUT2 have a role in intestinal glucose uptake? F1000Res. 2014 Dec 12;3:304. doi: 10.12688/f1000research.5934.1. eCollection 2014. PMID 25671087
- [Background] Naftalin RJ. A computer model simulating human glucose absorption and metabolism in health and metabolic disease states. F1000Res. 2016 Apr 12;5:647. doi: 10.12688/f1000research.8299.1. eCollection 2016. PMID 27347379
- [Background] Roder PV, Geillinger KE, Zietek TS, Thorens B, Koepsell H, Daniel H. The role of SGLT1 and GLUT2 in intestinal glucose transport and sensing. PLoS One. 2014 Feb 26;9(2):e89977. doi: 10.1371/journal.pone.0089977. eCollection 2014. PMID 24587162
- [Background] Russell M, Rees G, Benton D, Kingsley M. An exercise protocol that replicates soccer match-play. Int J Sports Med. 2011 Jul;32(7):511-8. doi: 10.1055/s-0031-1273742. Epub 2011 Apr 6. PMID 21472627
- [Background] Russell M, Benton D, Kingsley M. Influence of carbohydrate supplementation on skill performance during a soccer match simulation. J Sci Med Sport. 2012 Jul;15(4):348-54. doi: 10.1016/j.jsams.2011.12.006. Epub 2012 Jan 9. PMID 22230353
- [Background] Russell M, Benton D, Kingsley M. Carbohydrate ingestion before and during soccer match play and blood glucose and lactate concentrations. J Athl Train. 2014 Jul-Aug;49(4):447-53. doi: 10.4085/1062-6050-49.3.12. Epub 2014 Jun 16. PMID 24933430
- [Background] Russell M, Kingsley M. The efficacy of acute nutritional interventions on soccer skill performance. Sports Med. 2014 Jul;44(7):957-70. doi: 10.1007/s40279-014-0184-8. PMID 24728928
- [Background] Seidelmann SB, Feofanova E, Yu B, Franceschini N, Claggett B, Kuokkanen M, Puolijoki H, Ebeling T, Perola M, Salomaa V, Shah A, Coresh J, Selvin E, MacRae CA, Cheng S, Boerwinkle E, Solomon SD. Genetic Variants in SGLT1, Glucose Tolerance, and Cardiometabolic Risk. J Am Coll Cardiol. 2018 Oct 9;72(15):1763-1773. doi: 10.1016/j.jacc.2018.07.061. PMID 30286918
- [Background] Simulescu, V., Ilia, G., Macarie, L., & Merghes, P. (2019). Sport and energy drinks consumption before, during and after training. Science and Sports, 34(1), 3-9. https://doi.org/10.1016/j.scispo.2018.10.002
- [Background] Pfeiffer B, Stellingwerff T, Zaltas E, Jeukendrup AE. Oxidation of solid versus liquid CHO sources during exercise. Med Sci Sports Exerc. 2010 Nov;42(11):2030-7. doi: 10.1249/MSS.0b013e3181e0efc9. PMID 20404762
- [Background] Thazhath SS, Wu T, Young RL, Horowitz M, Rayner CK. Glucose absorption in small intestinal diseases. Expert Rev Gastroenterol Hepatol. 2014 Mar;8(3):301-12. doi: 10.1586/17474124.2014.887439. Epub 2014 Feb 6. PMID 24502537
- [Background] Thomas DT, Erdman KA, Burke LM. American College of Sports Medicine Joint Position Statement. Nutrition and Athletic Performance. Med Sci Sports Exerc. 2016 Mar;48(3):543-68. doi: 10.1249/MSS.0000000000000852. PMID 26891166
- [Background] Thorsen K, Drengstig T, Ruoff P. Transepithelial glucose transport and Na+/K+ homeostasis in enterocytes: an integrative model. Am J Physiol Cell Physiol. 2014 Aug 15;307(4):C320-37. doi: 10.1152/ajpcell.00068.2013. Epub 2014 Jun 4. PMID 24898586
- [Background] Scribbans TD, Vecsey S, Hankinson PB, Foster WS, Gurd BJ. The Effect of Training Intensity on VO2max in Young Healthy Adults: A Meta-Regression and Meta-Analysis. Int J Exerc Sci. 2016 Apr 1;9(2):230-247. doi: 10.70252/HHBR9374. eCollection 2016. PMID 27182424
- [Background] Zisko N, Stensvold D, Hordnes-Slagsvold K, Rognmo O, Nauman J, Wisloff U, Karlsen T. Effect of Change in VO2max on Daily Total Energy Expenditure in a Cohort of Norwegian Men: A Randomized Pilot Study. Open Cardiovasc Med J. 2015 Apr 30;9:50-7. doi: 10.2174/1874192401509010050. eCollection 2015. PMID 25969700